CLINICAL TRIAL: NCT06310590
Title: Study on the Safety and Effectiveness of NRT6003 Injection in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Safety and Efficacy of TareSphere in Patients With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu New Radiomedicine Technology Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRT6003-HCC-2022; CTR20230515 (Other: Center for Drug Evaluation, NMPA)
Record Dates: First submitted 2024-02-26; First posted 2024-03-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Selective internal radiation therapy; Yttrium-90; Transarterial Radioembolization;

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NRT6003 Injection (Experimental): Patients will be administered a single dose of NRT6003 Injection, and then they will be assessed by SPECT-CT imaging within 24 hours for its distribution in the chest and upper abdomen, including extrahepatic shunts, intrahepatic distribution, and target lesion distribution as expected.
  Nine Patients will be tested for the radioactivity of Yttrium-90 in blood, urine, and feces (if available).
  Interventions: Drug: NRT6003 Injection

INTERVENTIONS:
Drug: NRT6003 Injection — Selective internal radiation therapy (SIRT) with TareSphere
  Other Names: Yttrium-90 carbon microspheres

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of NRT6003 Injection in patients with unresectable HCC.

DETAILED DESCRIPTION:
The efficacy and safety of TareSphere in patients with unresectable HCC remains unknown. This trial is a prospective, multicenter, open-label, single-arm phase I trial designed to evaluate the safety and efficacy of NRT6003 injection.

The primary objective is to evaluate the safety of NRT6003 Injection. While the secondary objectives include the assessments of the antitumoral efficacy, the improvement of patients´ quality of life, and the distribution characteristics of Yttrium-90 in body.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 and signed informed consent;
2. Diagnosed as hepatocellular carcinoma clinically, by imaging and/or pathology based on the guideline of the National Health Commission of the People's Republic of China (2022);
3. Evaluated by the investigator as not suitable for surgical resection/ablation, or there are other reasons unsuitable for surgical resection/ablation, or the participant refuses surgical resection/ablation;
4. At least one well defined tumor (mRECIST), assessed by enhanced MRI or CT images;
5. Child-Pugh score ≤ 7;
6. Eastern Cooperative Oncology Group performance status ≤ 1;
7. Tumor burden ≤ 50 percent of the total liver volume;
8. Adequate organ function: (1) Blood routine [no blood transfusion or granulocyte colony-stimulating factor (G-CSF) treatment within 14 days]: absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet (PLT) ≥ 80 × 10^9/L; hemoglobin (HGB) ≥ 90 g/L; (2) Liver function: total bilirubin (TBIL) ≤ 2 times upper limit of normal (ULN); alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 5. 0×ULN; Albumin > 30 g/L; (3) Renal function: Creatinine (Cr) ≤ 1.5×ULN; creatinine clearance rate (CCr)≥ 50 mL/min (calculated according to Cockcroft-Gault formula); (4) Coagulation function: international normalized ratio (INR), prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN [If any participant takes warfarin or heparin for anticoagulation therapy, the investigator should evaluate whether the participant meet the requirements of the protocol]; (5) Cardiovascular function: left ventricular ejection fraction (LVEF) ≥ 50 percent assessed by ultrasonic cardiogram;
9. Women and men of childbearing age must agree to take strict and effective contraceptive measures during the study period and within 6 months after the end of the trial. Men are forbidden to donate sperm. The pregnancy test results of female participants of childbearing age during the screening period and within 24 hours before administration must be negative.

Exclusion Criteria:

1. With the extrahepatic metastasis or concurrent malignant tumors other than liver cancer;
2. With the hepatic tumor thrombus (excluding the thrombus limited to liver segments or lobes);
3. With hepatic artery malformation and unable to intubate hepatic artery;
4. Allergy to contrast agents or anesthetics;
5. Severe pulmonary dysfunction (forced expiratory volume in one second, FEV1/FVC < 50 percent or forced expiratory volume in one second (FEV1) < 50 percent of predicted value, or maximum voluntary ventilation (MVV) < 50 L/min);
6. With the clinical manifestations of decompensated liver cirrhosis (moderate or severe ascites, upper gastrointestinal bleeding, hepatic encephalopathy, etc.);
7. With diseases have not been controlled despite aggressive treatment, and which may affect the safety or the efficacy of the investigational drug in the judgement of investigators;
8. Active or severely infected participants requiring systemic therapy;
9. With positive results of HIV antibody test;
10. Estimated survival period < 3 months;
11. Have received radiotherapy or transcatheter arterial chemoembolization (participants who have received transcatheter arterial non-iodized oil chemoembolization are judged by investigators);
12. Technetium (99mTc)-macroaggregated albumin (MAA) hepatic arterial perfusion imaging estimates that the NRT6003 injection cannot cover all lesions within the liver (excluding lesions previously treated by the investigator as non-active or non-progressive);
13. Hepatic artery angiography and 99mTc-MAA hepatic artery perfusion imaging demonstrate gastrointestinal shunts, which may not be remedied through vascular intervention techniques;
14. 99mTc-MAA arterial perfusion imaging shows that the single lung radiation absorbed dose > 30 Gy;
15. Received antitumor therapy or participated in other interventional clinical trials within 30 days prior to dosing;
16. Pregnant or lactating women;
17. Have persistent, unrelieved toxicity reaction of CTCAE≥2 grade caused by previous antitumor treatment (excluding alopecia) judged by investigators;
18. Any other reason that the investigator deems the participant unsuitable for participating in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Adverse events/ Severe adverse events | Up to 12 months
  Occurrence of adverse events/severe adverse events
Localized Objective response rates (ORR) | Up to 6 months (initial tumor assessment after administration)
  Liver target lesions, evaluated based on the mRECIST criteria

SECONDARY OUTCOMES:
Hepatic time to progression (hTTP) | Up to 12 months
  Time to progression of liver target lesions, evaluated by the investigator and independent image review committee respectively (mRECIST)
Duration of response (DOR) | Up to 12 months
  Time without imaging progression, evaluated by the investigator and independent image review committee respectively (mRECIST)
Disease control rate (DCR) | Up to 12 months
  Time without imaging progression, evaluated by the investigator and independent image review committee respectively (mRECIST)
Time to progression (TTP) | Up to 12 months
  Time with tumor progression, evaluated by the investigator and independent image review committee respectively (mRECIST)
Progression Free Survival (PFS) | Up to 12 months
  Duration from the administration to the first evidence of progression or death from any cause, evaluated by the investigator and independent image review committee respectively (mRECIST)
Concentration of Alpha fetoprotein (AFP) | Up to 12 months
  The variation of AFP levels
Quality of life (QoL) | Up to 12 months
  The variation of QoL with the EORTC (European organization for Research and Treatment of Cancer) QLG (Quality of Life Group) Core Questionnaire (EORTC QLQ-C30)
Yttrium-90 distribution | Within 24 hours
  Assessed by SPECT-CT imaging in the chest and upper abdomen, including extrahepatic shunts, intrahepatic distribution, and target lesion distribution as expected.
Resection rate of liver target lesions | Within 6 months after administration
  Resection rate of liver target lesions
Radioactivity of Yttrium-90 for 9 participants, assessed by liquid scintillation counter | Within 168 hours
  Detect the radioactivity of Yttrium-90 in blood, urine, and feces (if available) in liquid scintillation counter

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (10):
- China (10):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No